CLINICAL TRIAL: NCT05120869
Title: Implementing Innovative and Strategic Approaches to Prevent and Mitigate the Deleterious Effects of HPV Across the Lifespan of Hispanics of Mexican Origin: Healthcare Provider Intervention
Brief Title: Healthcare Provider Human Papillomavirus Education and Professional Skills Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Burrell College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Eva Moya, Associate Professor, University of Texas, El Paso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 8321; 2U54MD007592-26 (NIH)
Record Dates: First submitted 2021-10-06; First posted 2021-11-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Health Personnel Attitude; Health Knowledge, Attitudes, Practice
Keywords: Healthcare Professionals; Health Personnel Knowledge, Attitudes, Practices; Healthcare Skills and Training; Human Papillomavirus Vaccination; Human Papillomavirus Cancer Screening; HPV Cancer Prevention; HPV Cancer Mitigation; Sexual and Reproductive Health; U.S.-Mexico Border Health; Behavioral Research; Community Engaged Research; Health Disparities; Health Inequities; Social Determinants of Health; Coronavirus disease 2019 (COVID-19) Pandemic
MeSH Terms: conditions — Behavior; Coitus; COVID-19

STUDY DESIGN:
Intervention Model Description: A parallel trial design will be used to examine the effectiveness of a tailored HPV education and professional skills intervention. Emerging and current healthcare providers will be randomly assigned to one of two conditions: 1) treatment condition in which they will receive a tailored Education and Professional Skills Intervention, and 2) control condition in which they will receive general, publicly available information about HPV and communication skills. Participants will then be followed over time and the responses will be compared between groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: * Participants [blinding]: participants will be randomly assigned to treatment and control groups, they will not be made aware of other participant's receipt of treatment or control materials. Participants will be asked not to discuss this project outside of the intervention; delivery of the intervention or other educational materials will be virtual, limiting the ability of participants to interact with one another during the study.
  * Outcome assessor [blinding]: to reduce bias in the implementation and assessment of the clinical trial, participant information and pre-post survey responses will be maintained separately from the assignment and delivery of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): A tailored HPV education and professional skills intervention.
  Interventions: Behavioral: Tailored HPV Education and Professional Skills Intervention Group
- Control (Active Comparator): General/publicly available educational materials on HPV and communication skills.
  Interventions: Behavioral: General HPV Education and Communication Skills Control Group

INTERVENTIONS:
Behavioral: Tailored HPV Education and Professional Skills Intervention Group — The provider education and professional skills intervention will involve audio and visual content and will be delivered in the English language.
  Arms: Treatment
Behavioral: General HPV Education and Communication Skills Control Group — The general provider education intervention will involve audio and visual content and will be delivered in the English language.
  Arms: Control

SUMMARY:
Healthcare providers (HCP) serving the El Paso U.S.-Mexico Border Region will be recruited to compare educational and professional skills interventions focused on the human papillomavirus (HPV). Our hypothesis is that improving provider knowledge and communication strategies about HPV and its vaccine will reduce hesitancy and increase uptake and completion among the populations they serve.

DETAILED DESCRIPTION:
A sample of emerging [in training] and current [in practice] health professionals from the El Paso U.S.-Mexico Border Region will be recruited to participate in a human papillomavirus (HPV) educational and professional skills intervention. Hypothesis: improving provider knowledge and communication strategies about HPV and its vaccine will reduce hesitancy and increase uptake and completion among eligible individuals through a tailored multi-media intervention to strengthen providers' ability to discuss HPV and vaccination in an informed and culturally competent manner, and increase subsequent provider recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Current (in practice) or emerging (in training - medical student, resident, or fellow) healthcare provider
* Working/training or living in the El Paso U.S.-Mexico Border Region (i.e., El Paso County, TX-Southern New Mexico)
* Have the authorization to recommend/prescribe/administer the HPV vaccine

Exclusion Criteria:

* Unaffiliated with the El Paso U.S.-Mexico Border Region (i.e., El Paso County, TX-Southern New Mexico)
* Participation in Phases I or II of the larger research project [cross-sectional phases]
* Does not identify as a current or emerging healthcare provider
* Declines or is unable to participate in the full intervention and follow-up time-points
* Unable to complete participation and activities in the English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Between-group changes in proportions from post-intervention scores of the Healthcare Provider (HCP) Practices scale on the Healthcare Personnel Survey | immediately post-intervention (0 months), 3 months post-intervention, and 6 months post-intervention
  8-item HCP Practices scale (HCP vaccine recommendations, HCP screening recommendations, HCP communication practices) scored on a Likert scale from Never (1) to Always (5)

SECONDARY OUTCOMES:
Between-group changes in proportions from post-intervention scores of the Human Papillomavirus (HPV) Vaccine Attitudes scale on the Healthcare Personnel Survey | immediately post-intervention (0 months), 3 months post-intervention, and 6 months post-intervention
  9-item HPV Vaccine Attitudes scale (perceived safety, perceived harm, perceived effectiveness) scored on a Likert scale from Strongly disagree (1) to Strongly agree (5)
Between-group changes in proportions from post-intervention scores on the Human Papillomavirus (HPV) Knowledge scale on the Healthcare Personnel Survey | immediately post-intervention (0 months), 3 months post-intervention, and 6 months post-intervention
  14-item HPV Knowledge scale scored as True (1) or False (0)

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Moya, PhD, LMSW, Principal Investigator — The University of Texas at El Paso, Border Biomedical Research Center
Locations (2):
- United States (2):
  - Burrell College of Osteopathic Medicine, Las Cruces, New Mexico
  - The University of Texas at El Paso, Border Biomedical Research Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Collected deidentified individual participant data (IPD), all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Approximately, starting 6 months-post scholarly publication of previously listed primary and secondary study outcome(s).
Access Criteria: Collected deidentified IPD and supporting information will be provided on a case by case basis following a formal request to the University of Texas at El Paso (UTEP) Institutional Review Board (IRB) and subsequent approval by the Principal Investigator.
URL: http://www.utep.edu/orsp/human-subjects-research/index.html

REFERENCES:
- [Background] Brabin L, Roberts SA, Farzaneh F, Kitchener HC. Future acceptance of adolescent human papillomavirus vaccination: a survey of parental attitudes. Vaccine. 2006 Apr 12;24(16):3087-94. doi: 10.1016/j.vaccine.2006.01.048. Epub 2006 Feb 9. PMID 16500736
- [Background] McRee AL, Brewer NT, Reiter PL, Gottlieb SL, Smith JS. The Carolina HPV immunization attitudes and beliefs scale (CHIAS): scale development and associations with intentions to vaccinate. Sex Transm Dis. 2010 Apr;37(4):234-9. doi: 10.1097/OLQ.0b013e3181c37e15. PMID 19940807
- [Background] Katz ML, Krieger JL, Roberto AJ. Human papillomavirus (HPV): college male's knowledge, perceived risk, sources of information, vaccine barriers and communication. J Mens Health. 2011 Oct 1;8(3):175-184. doi: 10.1016/j.jomh.2011.04.002. PMID 21966351
- [Derived] Martinez J, Cordero JI, Whitney M, LaRoche KL, Frietze G, Moya EM, Gosselink K. Web-Based Human Papillomavirus Education and Professional Skills Intervention for Health Care Providers: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 3;14:e60790. doi: 10.2196/60790. PMID 40179382
- See also: NIH RePORTER for 2U54MD007592-26 8321 — http://reporter.nih.gov/project-details/9828289